CLINICAL TRIAL: NCT02382913
Title: Phase 1 Extension Study to Evaluate Antibody Persistence Approximately 3 Years After Administration of Different Dosages of Acellular Pertussis or Tetanus-Diphtheria-acellular Pertussis Booster Vaccines in Healthy Adult Subjects Enrolled in Study V113_01
Brief Title: Persistency Study After aP / Tdap Booster Vaccines in Adult Subjects (V113_01 Extension 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: V113_01E1; 2014-003729-16 (EudraCT Number)
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group 1 (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: low dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart.
  Interventions: Biological: aP booster
- Group 2 (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: medium dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart.
  Interventions: Biological: aP booster
- Group 3 (Experimental): Subjects received acellular pertussis (aP) vaccine with different antigen dose formulations: high dose of PT, FHA, PRN, followed by one fixed dose of diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) administered one month apart
  Interventions: Biological: aP booster
- Group 4 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: low dose of PT, FHA, PRN, low dose of D (diphteria) toxoid, fixed dose of T (tetanus) toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: TdaP booster
- Group 5 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: medium dose of PT, FHA, PRN, low dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: TdaP booster
- Group 6 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: high dose of PT, FHA, PRN, low dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: TdaP booster
- Group 7 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: low dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: TdaP booster
- Group 8 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: medium dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart
  Interventions: Biological: TdaP booster
- Group 9 (Experimental): Subjects received tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) with different antigen dose formulations: high dose of PT, FHA, PRN, double dose of D toxoid, fixed dose of T toxoid, followed by one administration of saline solution one month apart.
  Interventions: Biological: TdaP booster
- Group 10 (Active Comparator): Subject received one dose of a licensed TdaP booster vaccine (containing 8 μg each of PT, FHA and 2.5 μg of PRN antigens and 2.5 Lf of diphtheria toxoid and 5 Lf of tetanus toxoid) followed by one administration of saline solution one month apart
  Interventions: Biological: Licensed TdaP booster (Boostrix®)

INTERVENTIONS:
Biological: aP booster — Acellular pertussis vaccine:
  Acellular pertussis (aP) vaccine was administered with different antigen doses intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Biological: Diphtheria and tetanus vaccine (adsorbed, reduced antigen content, Germany) To ensure all subjects receive a tetanus and diphtheria booster vaccination, an injection was administered on Study Day 30, one month after the administration of the investigational vaccine.
  Arms: Group 1; Group 2; Group 3
Biological: TdaP booster — Tetanus, reduced diphtheria, and acellular pertussis vaccine (adsorbed) Tetanus, reduced diphtheria, and acellular pertussis (TdaP) vaccine was administered with different antigen doses intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Other: Saline solution Subjects received one injection of saline solution at one month after vaccination.
  Arms: Group 4; Group 5; Group 6; Group 7; Group 8; Group 9
Biological: Licensed TdaP booster (Boostrix®) — Licensed TdaP booster vaccine Licenced TdaP booster vaccine was administered intramuscularly in the upper deltoid region of the subject's non-dominant arm.
  Other: Saline solution Subjects received one injection of saline solution at one month after vaccination.
  Arms: Group 10

SUMMARY:
The purpose of this study is to evaluate the persistence of immune response against the three pertussis antigens (anti- pertussis toxoid (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN)) in subjects who received a booster dose of either aP or Tdap study vaccines or Boostrix® during V113_01 study.

There was only one Clinic Visit at day 1. Eligible subjects went undergo a single blood draw after which they were observed for approximately 15 minutes. Approximately 10.0 mL of blood was withdrawn.

No vaccine was administered and no safety data was collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals previously enrolled in V113_01 trial, who completed the study following study protocol and who received the appropriate booster vaccine per group assignment
* Individuals who voluntarily gave written informed consent after the nature of the study was explained according to local regulatory requirements, prior to study entry
* Individuals who could comply with study procedures including follow-up

Exclusion Criteria:

1. Clinical conditions representing a contraindication to blood draw.
2. Abnormal function of the immune system resulting from:

   * Clinical conditions
   * Systemic administration of corticosteroids per oral (PO)/ intravenous (IV)/ intramuscular (IM) for more than 14 consecutive days within 90 days prior to informed consent.
   * Administration of antineoplastic and immunomodulating agents or radiotherapy within 90 days prior to informed consent.
3. Received immunoglobulins or any blood products within 180 days prior to informed consent.
4. Received an investigational or non-registered medicinal product within 30 days prior to informed consent
5. Study personnel as an immediate family or household member
6. Any other clinical condition that, in the opinion of the investigator, could interfere with the results of the study or pose additional risk to the subject due to participation in the study

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 315 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 02, Center for Vaccinology (CEVAC), Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Leroux-Roels G, Lattanzi M, Solis CD, Contorni M, Costantini M, Moraschini L, Bardelli M, Bertholet S, Borgogni E, Buricchi F, Cantisani R, Faenzi E, Finco O, Leuzzi R, Pizza M, Rosa D, Schiavetti F, Seubert A, Spensieri F, Volpini G, Zedda L, Giudice GD, Galgani I. A phase I, randomized, controlled, dose-ranging study of investigational acellular pertussis (aP) and reduced tetanus-diphtheria-acellular pertussis (TdaP) booster vaccines in adults. Hum Vaccin Immunother. 2018 Jan 2;14(1):45-58. doi: 10.1080/21645515.2017.1385686. Epub 2017 Nov 27. PMID 29172945

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one site in Belgium.
  - V113_01 parent study number: NCT01529645
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Group aP1: Subjects received a single dose of aP booster vaccine (containing a low dose of PT, FHA and PRN antigens) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group aP2: Subjects received a single dose of aP booster vaccine (containing a medium dose of PT, FHA and PRN antigens) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group aP4: Subjects received a single dose of aP booster vaccine (containing a high dose of PT, FHA and PRN antigens) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D2aP1: Subjects received a single dose of TdaP booster vaccine (containing a low dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D2aP2: Subjects received a single dose of TdaP booster vaccine (containing a medium dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D2aP4: Subjects received a single dose of TdaP booster vaccine (containing a high dose of PT, FHA, PRN antigens, a low dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D4aP1: Subjects received a single dose of TdaP booster vaccine (containing a low dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D4aP2: Subjects received a single dose of TdaP booster vaccine (containing a medium dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Group T5D4aP4: Subjects received a single dose of TdaP booster vaccine (containing a high dose of PT, FHA, PRN antigens, a double dose of diphtheria toxoid and a fixed dose of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
- Licensed Tdap: Subjects received a single dose of a comparator TdaP booster vaccine (containing 8 μg each of PT, FHA and 2.5 μg of PRN antigens and 2.5 Lf of diphtheria toxoid and 5 Lf of tetanus toxoid) on parent study V113_01 and had blood collected at approximately 3 years later, in current V113_01E1 study.
Period: Overall Study
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed Tdap
Started | 27 | 36 | 32 | 27 | 33 | 30 | 37 | 30 | 30 | 33
Completed | 27 | 36 | 32 | 27 | 33 | 30 | 37 | 30 | 30 | 33
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed Tdap | Total
Number analyzed (Participants) | 27 | 36 | 32 | 27 | 33 | 30 | 37 | 30 | 30 | 33 | 315
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.7) | 29.5 (4.9) | 30.3 (6.4) | 31.3 (6.3) | 30.9 (5.7) | 30 (5.6) | 28.2 (4.4) | 30.1 (4.6) | 31.3 (5.9) | 31.5 (6.7) | 30.3 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 25 | 19 | 11 | 19 | 16 | 27 | 13 | 19 | 21 | 187
  Male | 10 | 11 | 13 | 16 | 14 | 14 | 10 | 17 | 11 | 12 | 128

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in aP1, aP2, aP4 Groups Against Pertussis Antigens at Day 1.
Description: The antibody response against the pertussis antigen components (PT, FHA and PRN) at day 1 as measured by Multiplex ELISA and reported as Geometric Mean Concentrations (GMCs) in aP1, aP2, aP4 Groups versus the response to the commercially available Tdap comparator.
  Note: The mean and confidence intervals of Licensed Tdap for the same antigen can be different (from aP to Tdap table) since two different statistical model were fitted within each antigen: one with aP and Licensed Tdap groups and one with Tdap and Licensed Tdap groups.
Time Frame: Day 1
Population: Analysis were done on per protocol set (PPS) i.e., All subjects in the all enrolled set who provided immunogenicity data at V113_01E1 visit 1 and:
  * correctly received the vaccine in the V113_01 parent study
  * had no major protocol deviations leading to exclusion or were not excluded due to other reasons as defined prior to analysis
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Licensed Tdap
Number analyzed (Participants) | 27 | 34 | 32 | 32
IU/mL
  PT | 28 [18 to 44] | 31 [21 to 46] | 48 [32 to 72] | 18 [12 to 27]
  FHA | 43 [31 to 59] | 54 [41 to 71] | 60 [45 to 80] | 63 [47 to 84]
  PRN | 206 [138 to 308] | 276 [193 to 394] | 396 [274 to 572] | 126 [87 to 182]

2. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in T5D2aP1, T5D2aP2 and T5D2aP4 Groups Against Pertussis Antigens at Day 1.
Description: The antibody response against the pertussis antigen components (PT, FHA and PRN) in serum at day 1 as measured by Multiplex ELISA and reported as Geometric Mean Concentrations (GMCs) in T5D2aP1, T5D2aP2 and T5D2aP4 Groups versus the response to the commercially available Tdap comparator.
  Note: The mean and confidence intervals of Licensed Tdap for the same antigen can be different (from aP to Tdap table) since two different statistical model were fitted within each antigen: one with aP and Licensed Tdap groups and one with Tdap and Licensed Tdap groups.
Time Frame: Day 1
Population: Analysis were done on per protocol set.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Licensed Tdap
Number analyzed (Participants) | 26 | 31 | 28 | 32
IU/mL
  PT | 17 [12 to 24] | 22 [15 to 31] | 34 [24 to 48] | 18 [13 to 25]
  FHA | 41 [29 to 56] | 32 [24 to 44] | 51 [37 to 69] | 63 [47 to 84]
  PRN | 93 [59 to 146] | 248 [165 to 375] | 373 [242 to 575] | 126 [84 to 189]

3. Primary Outcome: Geometric Mean Concentrations (GMCs) of Antibodies in T5D4aP1, T5D4aP2 and T5D4aP4 Groups Against Pertussis Antigens at Day 1.
Description: The antibody response against the pertussis antigen components (PT, FHA and PRN) in serum at day 1 as measured by Multiplex ELISA and reported as Geometric Mean Concentrations (GMCs) in T5D4aP1, T5D4aP2 and T5D4aP4 Groups versus the response to the commercially available Tdap comparator.
  Note: The mean and confidence intervals of Licensed Tdap for the same antigen can be different (from aP to Tdap table) since two different statistical model were fitted within each antigen: one with aP and Licensed Tdap groups and one with Tdap and Licensed Tdap groups.
Time Frame: Day 1
Population: Analysis were done on per protocol set.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed Tdap
Number analyzed (Participants) | 33 | 28 | 29 | 32
IU/mL
  PT | 31 [22 to 43] | 31 [21 to 44] | 43 [30 to 61] | 18 [13 to 25]
  FHA | 51 [38 to 67] | 48 [35 to 65] | 58 [43 to 78] | 63 [47 to 84]
  PRN | 247 [166 to 368] | 266 [172 to 410] | 292 [191 to 448] | 126 [84 to 189]

4. Primary Outcome: Geometric Mean Ratios Antibodies Concentrations in aP1, aP2, aP4 Groups as Measured at V113_01E1 Day 1 vs. All V113_01 Time Points.
Description: Geometric Mean Ratios of anti-PT, anti-FHA and anti-PRN antibody were calculated to measure the changes in immunogenicity concentrations within subjects from all V113_01 time points to V113_01E1 day 1.
  Note: The mean and confidence intervals of Licensed Tdap for the same antigen can be different (from aP to Tdap table) since two different statistical model were fitted within each antigen: one with aP and Licensed Tdap groups and one with Tdap and Licensed Tdap groups.
Time Frame: Day 1, Day 8, Day 30, Day 180, Day 365 of V113_01 and Day 1 of V113_01E1
Population: Analysis were done on per protocol set. Note: Number of participants analyzed for Day 1 of V113_01E1/ Day 180 of V113_01 PT, FHA and PRN was 27, 32, 31, 32 respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Licensed Tdap
Number analyzed (Participants) | 27 | 34 | 32 | 32
Ratios
  Day 1 of V113_01E1/ Day 1 of V113_01 (PT) | 7.21 [4.77 to 11] | 7.63 [5.29 to 11] | 11 [7.48 to 16] | 4.28 [2.93 to 6.25]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PT) | 2.93 [1.83 to 4.69] | 1.50 [0.99 to 2.28] | 1.60 [1.04 to 2.46] | 1.00 [0.65 to 1.54]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PT) | 0.30 [0.24 to 0.38] | 0.24 [0.20 to 0.30] | 0.26 [0.21 to 0.32] | 0.21 [0.17 to 0.26]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PT) | 0.48 [0.41 to 0.56] | 0.45 [0.39 to 0.52] | 0.42 [0.36 to 0.48] | 0.42 [0.36 to 0.49]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PT) | 0.68 [0.59 to 0.79] | 0.63 [0.55 to 0.72] | 0.56 [0.49 to 0.64] | 0.67 [0.59 to 0.77]
  Day 1 of V113_01E1/ Day 1 of V113_01 (FHA) | 2.25 [1.67 to 3.05] | 3.25 [2.49 to 4.25] | 2.75 [2.09 to 3.63] | 3.36 [2.55 to 4.44]
  Day 1 of V113_01E1/ Day 8 of V113_01 (FHA) | 1.06 [0.77 to 1.46] | 1.00 [0.75 to 1.32] | 0.93 [0.69 to 1.24] | 0.62 [0.46 to 0.83]
  Day 1 of V113_01E1/ Day 30 of V113_01 (FHA) | 0.39 [0.30 to 0.50] | 0.34 [0.27 to 0.43] | 0.32 [0.25 to 0.40] | 0.26 [0.21 to 0.33]
  Day 1 of V113_01E1/ Day 180 of V113_01 (FHA) | 0.64 [0.54 to 0.77] | 0.69 [0.58 to 0.81] | 0.65 [0.55 to 0.77] | 0.54 [0.45 to 0.63]
  Day 1 of V113_01E1/ Day 365 of V113_01 (FHA) | 0.83 [0.70 to 0.98] | 0.95 [0.82 to 1.10] | 0.78 [0.67 to 0.91] | 0.79 [0.68 to 0.92]
  Day 1 of V113_01E1/ Day 1 of V113_01 (PRN) | 11 [6.75 to 17] | 15 [10 to 23] | 20 [13 to 31] | 6.61 [4.36 to 10]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PRN) | 1.66 [1.12 to 2.45] | 1.31 [0.92 to 1.85] | 0.85 [0.59 to 1.22] | 0.88 [0.61 to 1.26]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PRN) | 0.33 [0.26 to 0.41] | 0.30 [0.24 to 0.36] | 0.27 [0.22 to 0.33] | 0.29 [0.24 to 0.36]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PRN) | 0.45 [0.39 to 0.51] | 0.47 [0.42 to 0.54] | 0.47 [0.42 to 0.54] | 0.48 [0.42 to 0.54]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PRN) | 0.62 [0.55 to 0.70] | 0.63 [0.56 to 0.70] | 0.59 [0.53 to 0.66] | 0.72 [0.64 to 0.80]

5. Primary Outcome: Geometric Mean Ratios Antibodies Concentrations in T5D2aP1, T5D2aP2 and T5D2aP4 Groups as Measured at V113_01E1 Day 1 vs. All V113_01 Time Points.
Description: as for outcome 4
Time Frame: Day 1, Day 8, Day 30, Day 180, Day 365 of V113_01 and Day 1 of V113_01E1
Population: Analysis were done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Licensed Tdap
Number analyzed (Participants) | 26 | 31 | 28 | 32
Ratios
  Day 1 of V113_01E1/ Day 1 of V113_01 (PT) | 3.70 [2.40 to 5.71] | 3.58 [2.41 to 5.32] | 6.67 [4.39 to 10] | 4.28 [2.90 to 6.33]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PT) | 1.05 [0.71 to 1.55] | 1.03 [0.72 to 1.46] | 0.80 [0.55 to 1.16] | 1.00 [0.71 to 1.42]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PT) | 0.30 [0.24 to 0.37] | 0.30 [0.25 to 0.36] | 0.26 [0.21 to 0.32] | 0.21 [0.17 to 0.25]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PT) | 0.44 [0.37 to 0.52] | 0.47 [0.40 to 0.56] | 0.41 [0.35 to 0.49] | 0.42 [0.36 to 0.49]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PT) | 0.70 [0.61 to 0.81] | 0.63 [0.56 to 0.72] | 0.61 [0.53 to 0.70] | 0.67 [0.59 to 0.77]
  Day 1 of V113_01E1/ Day 1 of V113_01 (FHA) | 1.99 [1.46 to 2.71] | 1.79 [1.35 to 2.39] | 2.04 [1.51 to 2.75] | 3.36 [2.54 to 4.45]
  Day 1 of V113_01E1/ Day 8 of V113_01 (FHA) | 0.94 [0.71 to 1.24] | 0.78 [0.60 to 1.00] | 0.84 [0.64 to 1.09] | 0.62 [0.48 to 0.79]
  Day 1 of V113_01E1/ Day 30 of V113_01 (FHA) | 0.49 [0.37 to 0.64] | 0.39 [0.31 to 0.51] | 0.40 [0.31 to 0.52] | 0.26 [0.21 to 0.34]
  Day 1 of V113_01E1/ Day 180 of V113_01 (FHA) | 0.76 [0.62 to 0.94] | 0.63 [0.52 to 0.77] | 0.66 [0.54 to 0.81] | 0.54 [0.44 to 0.65]
  Day 1 of V113_01E1/ Day 365 of V113_01 (FHA) | 0.94 [0.77 to 1.13] | 0.84 [0.70 to 1.00] | 0.87 [0.72 to 1.05] | 0.79 [0.67 to 0.94]
  Day 1 of V113_01E1/ Day 1 of V113_01 (PRN) | 7.65 [4.71 to 12] | 10 [6.71 to 16] | 11 [6.91 to 18] | 6.61 [4.27 to 10]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PRN) | 1.41 [0.96 to 2.06] | 1.11 [0.78 to 1.57] | 0.91 [0.63 to 1.32] | 0.88 [0.62 to 1.24]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PRN) | 0.35 [0.28 to 0.43] | 0.32 [0.26 to 0.39] | 0.30 [0.24 to 0.37] | 0.29 [0.24 to 0.36]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PRN) | 0.43 [0.36 to 0.50] | 0.47 [0.41 to 0.55] | 0.50 [0.43 to 0.59] | 0.48 [0.41 to 0.55]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PRN) | 0.70 [0.62 to 0.79] | 0.60 [0.54 to 0.73] | 0.59 [0.52 to 0.67] | 0.72 [0.64 to 0.80]

6. Primary Outcome: Geometric Mean Ratios Antibodies Concentrations in T5D4aP1, T5D4aP2 and T5D4aP4 Groups as Measured at V113_01E1 Day 1 vs. All V113_01 Time Points.
Description: as for outcome 4
Time Frame: Day 1, Day 8, Day 30, Day 180, Day 365 of V113_01 and Day 1 of V113_01E1
Population: Analysis were done on per protocol set. Note: Number of participants analyzed for Day 1 of V113_01E1/ Day 180 of V113_01 FHA and PRN was 33, 28, 28, 32 respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratios
Arm/Group | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed Tdap
Number analyzed (Participants) | 33 | 28 | 29 | 32
Ratios
  Day 1 of V113_01E1/ Day 1 of V113_01 (PT) | 3.40 [2.32 to 5.00] | 3.82 [2.51 to 5.79] | 5.90 [3.92 to 8.90] | 4.28 [2.90 to 6.33]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PT) | 1.02 [0.73 to 1.44] | 0.98 [0.67 to 1.42] | 1.11 [0.77 to 1.60] | 1.00 [0.71 to 1.42]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PT) | 0.37 [0.30 to 0.45] | 0.32 [0.26 to 0.39] | 0.32 [0.26 to 0.39] | 0.21 [0.17 to 0.25]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PT) | 0.60 [0.52 to 0.71] | 0.44 [0.37 to 0.53] | 0.48 [0.40 to 0.57] | 0.42 [0.36 to 0.49]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PT) | 0.81 [0.71 to 0.92] | 0.64 [0.56 to 0.73] | 0.65 [0.57 to 0.74] | 0.67 [0.59 to 0.77]
  Day 1 of V113_01E1/ Day 1 of V113_01 (FHA) | 2.09 [1.58 to 2.75] | 1.67 [1.23 to 2.25] | 2.19 [1.63 to 2.94] | 3.36 [2.54 to 4.45]
  Day 1 of V113_01E1/ Day 8 of V113_01 (FHA) | 0.85 [0.67 to 1.09] | 0.82 [0.63 to 1.08] | 0.99 [0.76 to 1.28] | 0.62 [0.48 to 0.79]
  Day 1 of V113_01E1/ Day 30 of V113_01 (FHA) | 0.45 [0.36 to 0.58] | 0.49 [0.38 to 0.64] | 0.50 [0.39 to 0.65] | 0.26 [0.21 to 0.34]
  Day 1 of V113_01E1/ Day 180 of V113_01 (FHA) | 0.78 [0.65 to 0.95] | 0.72 [0.58 to 0.88] | 0.79 [0.64 to 0.97] | 0.54 [0.44 to 0.65]
  Day 1 of V113_01E1/ Day 365 of V113_01 (FHA) | 0.99 [0.84 to 1.18] | 0.83 [0.69 to 1.00] | 0.97 [0.81 to 1.17] | 0.79 [0.67 to 0.94]
  Day 1 of V113_01E1/ Day 1 of V113_01 (PRN) | 8.76 [5.70 to 13] | 12 [7.50 to 19] | 13 [8.23 to 21] | 6.61 [4.27 to 10]
  Day 1 of V113_01E1/ Day 8 of V113_01 (PRN) | 1.24 [0.88 to 1.73] | 1.41 [0.98 to 2.03] | 1.11 [0.77 to 1.59] | 0.88 [0.62 to 1.24]
  Day 1 of V113_01E1/ Day 30 of V113_01 (PRN) | 0.33 [0.27 to 0.40] | 0.37 [0.30 to 0.46] | 0.33 [0.27 to 0.40] | 0.29 [0.24 to 0.36]
  Day 1 of V113_01E1/ Day 180 of V113_01 (PRN) | 0.57 [0.49 to 0.66] | 0.49 [0.41 to 0.57] | 0.48 [0.41 to 0.56] | 0.48 [0.41 to 0.55]
  Day 1 of V113_01E1/ Day 365 of V113_01 (PRN) | 0.67 [0.60 to 0.75] | 0.64 [0.57 to 0.73] | 0.58 [0.52 to 0.66] | 0.72 [0.64 to 0.80]

ADVERSE EVENTS:
Time Frame: No Adverse Events data were collected in this study.
Arm/Group | Group aP1 | Group aP2 | Group aP4 | Group T5D2aP1 | Group T5D2aP2 | Group T5D2aP4 | Group T5D4aP1 | Group T5D4aP2 | Group T5D4aP4 | Licensed Tdap
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.